CLINICAL TRIAL: NCT05768854
Title: An Open-label, Randomized, Active-Controlled, Phase 3 Study of Setrusumab Compared With Bisphosphonates in Pediatric Subjects With Osteogenesis Imperfecta Types I, III or IV
Brief Title: Setrusumab vs Bisphosphonates in Pediatric Subjects With Osteogenesis Imperfecta
Acronym: Cosmic
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UX143-CL314; 2023-504196-24-00 (Other: EU CT Number)
Record Dates: First submitted 2023-03-03; First posted 2023-03-14 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Diphosphonates; setrusumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous Bisphosphonates (IV-BP) -> Setrusumab (Active Comparator): Participants on IV-BP will continue their existing dose/regimen per investigator discretion; for participants not on IV-BP, the dose/regimen will be determined by the investigator.
  After the active-controlled period, participants will receive Setrusumab during the extension period
  Interventions: Drug: Bisphosphonate; Biological: Setrusumab
- Setrusumab (Experimental): Participants will receive Setrusumab during the active-controlled and extension period
  Interventions: Biological: Setrusumab

INTERVENTIONS:
Drug: Bisphosphonate — Administered per investigator discretion via intravenous (IV) infusion
  Arms: Intravenous Bisphosphonates (IV-BP) -> Setrusumab
Biological: Setrusumab — A fully human sclerostin neutralizing monoclonal antibody (mAb) administered once a month (QM) via intravenous (IV) infusion
  Other Names: BPS804; UX143

SUMMARY:
The primary objective of the study is to evaluate the effect of setrusumab vs intravenous bisphosphonates (IV-BP) on reduction in fracture rate, including morphometric vertebral fractures in pediatric participants.

DETAILED DESCRIPTION:
Participants will be randomized 1:1 to receive either setrusumab or IV-BP. Following randomization, participants will receive setrusumab or IV-BP for up to 24 months during the Active-controlled Period. At the end of the Active-controlled Period all participants will enter the Extension Period and participants assigned to IV-BP will transition to setrusumab. During the Extension Period, all participants will receive setrusumab for a minimum of 12 months or until setrusumab becomes commercially available in their respective country or the study is discontinued. The use of any bisphosphonate is prohibited throughout the Extension Period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 2 to < 7 years of age at time of informed consent
* Clinical diagnosis of OI Types I, III, or IV confirmed by identification of genetic mutation in COL1A1 or COL1A2
* History of ≥ 1 fracture in the past 12 months, ≥ 2 fractures in the past 24 months, or ≥ 1 femur, tibia, or humerus fracture in the past 24 months
* Any prior exposure to, or currently receiving, IV-bisphosphonate therapy for treatment of OI
* Serum 25-hydroxyvitamin D level ≥ 20 ng/mL at the Screening visit. If 25-hydroxyvitamin D levels are below 20 ng/mL, the subject may be rescreened after a minimum of 14 days of vitamin D supplementation as directed by the Investigator

Exclusion Criteria:

* Contraindication for the use of IV bisphosphonates based on clinical judgment of the Investigator
* History of skeletal malignancies or bone metastases at any time
* History of neural foraminal stenosis (except if due to scoliosis)
* Clinical manifestations of Chiari malformation or basilar invagination. Presence of any other neurologic disease that has been clinically unstable within past 2 years requires review by the Medical Monitor.
* History of or current uncontrolled concomitant diseases that may impact bone metabolism, such as hypo/hyperparathyroidism, abnormal thyroid function, nephrotic syndrome, or Stage IV/V renal disease
* Any skeletal condition (other than OI) leading to bone deformity and/or increased risk of fractures, such as rickets, osteopetrosis, idiopathic juvenile osteoporosis, or skeletal dysplasia
* History of known cardiovascular disease such as coronary artery anomaly, Kawasaki disease, myocarditis, cardiomyopathy, myocardial infarction, stroke, or thromboembolic disease. Individuals with other congenital or acquired cardiovascular disease necessitating echocardiogram require Medical Monitor review. Investigators should consider whether the potential benefits of treatment outweigh the potential risks in patients with cardiovascular risk factors such as confirmed arterial hypertension.
* Hypocalcemia, defined as serum calcium levels below the age-adjusted normal limit reference ranges after a recommended ≥ 4 hour fast, at Screening
* Estimated glomerular filtration rate <=35 mL/min/1.73 m2 at Screening
* Prior treatment with growth hormone, denosumab, anti-sclerostin antibody, or other anabolic or anti-resorptive medications impacting the bone (other than bisphosphonates) at any time
* History of external radiation therapy
* Known hypersensitivity to setrusumab or its excipients that, in the judgment of the Investigator, places the subject at increased risk for adverse effects
* Presence or history of any condition that, in the view of the Investigator, would interfere with participation, pose undue risk, or would confound interpretation of results
* Use of any investigational product or investigational medical device within 4 weeks or 5 half-lives (whichever is longer) of investigational drug prior to Screening, or during the study (per discretion of the Investigator in consultation with the Medical Monitor)
* Concurrent participation in another clinical study without prior approval from the study Medical Monitor

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Annualized Rate of All Radiographically-Confirmed Fractures, Including Morphometric Vertebral Fractures, at the Primary Analysis | Up to 24 Months

SECONDARY OUTCOMES:
Annualized Rate of Radiographically-Confirmed Fractures, Excluding Morphometric Vertebral Fractures, but Including Fractures of the Fingers, Toes, Face and Skull at the Primary Analysis | Up to 24 Months
Annualized Rate of All Radiographically-Confirmed Fractures, Excluding Morphometric Vertebral Fractures, and Fractures of the Fingers, Toes, Face and Skull, at the Primary Analysis | Up to 24 Months
Change from Baseline in Dual-energy X-ray Absorptiometry (DXA) Bone Mineral Density (BMD) Z-score at the Lumbar Spine at the Primary Analysis | Up to 24 Months
Proportion of Participants Experiencing New Radiographically-Confirmed Fractures, including Morphometric Vertebral Fractures, at the Primary Analysis | Up to 24 Months
Change from Baseline in Pediatric Orthopedic Society of North America Pediatric Outcomes Data Collection Instrument (POSNA-PODCI) Sports/Physical Functioning and Pain/Comfort Subscale Scores at the Primary Analysis | Baseline, Up to 24 Months
Percent Change from Baseline in DXA BMD at the Lumbar Spine at the Primary Analysis | Up to 24 Months
Serum Setrusumab Concentration | Up to 24 Months
Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) | Up to 24 Months
Number of Participants With Anti-Setrusumab Binding and Neutralizing Antibodies | Up to 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (20):
- United States (13):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Childrens Hospital LA, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Nemours/ Alfred i. duPoint Hospital for Children, Wilmington, Delaware
  - Children's National Hospital DC, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Shriners Hospitals for Children Chicago, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - University of North Carolina at Chapel Hill (UNC), Chapel Hill, North Carolina
  - Vanderbilt University Medical Center (VUMC), Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
- Hospital de Clinicas de Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil
- Canada (2):
  - Children's Hospital at London Health Sciences Centre, London, Ontario
  - Childrens Hospital Of Eastern Ontario Research Institute, University Of Ottawa, Ottawa
- Institut Imagine, Paris, France
- Azienda Ospedaliera Universitaria Policlinico Umberto I, Roma, Italy
- Universitair Medisch Centrum Utrecht (UMCU) - Wilhelmina Kinderziekenhuis, Utrecht, Netherlands
- Uniwersytet Medyczny w Lodzi - Klinika Endokrynologii i Chorob Metabolicznych, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Osteogenesis Imperfecta (OI) Research Study — https://www.ultraclinicaltrials.com/OI
- See also: Ultragenyx Transparency Commitment — https://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/